CLINICAL TRIAL: NCT01559116
Title: Randomised, Double-blind, Placebo-controlled, 6 Treatment, 4 Period, Incomplete Cross-over Trial to Characterise the 24-hour Lung Function Profiles of Tiotropium + Olodaterol Fixed Dose Combination (2.5/5 µg, 5/5 µg), Tiotropium (2.5 µg, 5 µg) and Olodaterol (5 µg) (Oral Inhalation, Delivered by the Respimat® Inhaler) After 6 Weeks Once Daily Treatment in Patients With Chronic Obstructive Pulmonary Disease (COPD) [VIVACITOTM]
Brief Title: Characterization of 24-hour Lung Function Profiles of Inhaled Tiotropium + Olodaterol Fixed Dose Combination in Patients Suffering From Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.20; 2011-004710-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; Tiotropium Bromide; olodaterol

ARMS (6):
- tiotropium+olodaterol FDC low dose (Experimental): tiotropium+olodaterol FDC low dose; 2 inhalations once daily (a.m. dosing)
  Interventions: Drug: tiotropium + olodaterol; Device: Respimat
- tiotropium+olodaterol FDC high dose (Experimental): tiotropium+olodaterol FDC high dose; 2 inhalations once daily (a.m. dosing)
  Interventions: Drug: tiotropium + olodaterol; Device: Respimat
- tiotropium low dose (Active Comparator): tiotropium low dose; 2 inhalations once daily (a.m. dosing)
  Interventions: Drug: tiotropium; Device: Respimat
- tiotropium high dose (Active Comparator): tiotropium high dose; 2 inhalations once daily (a.m. dosing)
  Interventions: Drug: tiotropium; Device: Respimat
- olodaterol (Active Comparator): one dose only; 2 inhalations once daily (a.m. dosing)
  Interventions: Drug: olodaterol; Device: Respimat
- placebo (Placebo Comparator): 2 inhalations once daily (a.m. dosing)
  Interventions: Drug: Placebo; Device: Respimat

INTERVENTIONS:
Drug: tiotropium + olodaterol — low dose + one dose only
  Arms: tiotropium+olodaterol FDC high dose
Drug: tiotropium — low dose
  Arms: tiotropium low dose
Drug: olodaterol — one dose only
  Arms: olodaterol
Drug: tiotropium — high dose
  Arms: tiotropium high dose
Drug: tiotropium + olodaterol — low dose + one dose only
  Arms: tiotropium+olodaterol FDC low dose
Drug: Placebo — placebo matching tiotropium+olodaterol FDC
  Arms: placebo
Device: Respimat — Respimat inhaler

SUMMARY:
The primary objective of the trial is to determine the 24-hour FEV1-time profile of tiotropium + olodaterol FDC, administered once daily by the RESPIMAT Inhaler after 6 weeks of treatment.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of chronic obstructive pulmonary disease
2. Relatively stable airway obstruction with a post-bronchodilator FEV1< 80% of predicted normal and a post-bronchodilator FEV1/FVC <70%
3. Male or female patients, 40 years of age or older
4. Smoking history of more than 10 pack years
5. Ability to perform technically acceptable pulmonary function tests and maintain records
6. Ability to inhale medication in a competent manner from the RESPIMAT Inhaler and from a metered dose inhaler (MDI)

Exclusion criteria:

1. significant disease other than COPD
2. clinically relevant abnormal lab values
3. history of asthma
4. diagnosis of thyrotoxicosis
5. diagnosis of paroxysmal tachycardia
6. history of myocardial infarction
7. unstable or life-threatening cardiac arrhythmia
8. Hospitalization for heart failure within the past year
9. known active tuberculosis
10. malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
11. history of life-threatening pulmonary obstruction
12. history of cystic fibrosis
13. clinically evident bronchiectasis
14. history of significant alcohol or drug abuse
15. history of thoracotomy with pulmonary resection
16. oral or patch ß-adrenergics
17. oral corticosteroid medication at unstable doses
18. regular use daytime oxygen therapy for more than one hour per day
19. Pulmonary rehabilitation program in the six weeks prior to the screening visit
20. Investigational drug within one month or six half lives (whichever is greater) prior to screening visit
21. Known hypersensitivity to ß-adrenergic drugs, BAC, EDTA
22. Pregnant or nursing women
23. Women of childbearing potential not using a highly effective method of birth control
24. Patients who have previously been randomised in this study or are currently participating in another study
25. Patients who are unable to comply with pulmonary medication restrictions prior to randomisation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (29):
- United States (4):
  - 1237.20.1204 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1237.20.1203 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1237.20.1201 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.20.1202 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
- Belgium (3):
  - 1237.20.32203 Boehringer Ingelheim Investigational Site, Genk
  - 1237.20.32201 Boehringer Ingelheim Investigational Site, Ghent
  - 1237.20.32204 Boehringer Ingelheim Investigational Site, Jambes
- Canada (2):
  - 1237.20.02202 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1237.20.02201 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Denmark (3):
  - 1237.20.45002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1237.20.45003 Boehringer Ingelheim Investigational Site, Odense C
  - 1237.20.45001 Boehringer Ingelheim Investigational Site, Silkeborg
- Germany (7):
  - 1237.20.49205 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.20.49204 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1237.20.49203 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.20.49206 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.20.49201 Boehringer Ingelheim Investigational Site, Mannheim
  - 1237.20.49207 Boehringer Ingelheim Investigational Site, Mönchengladbach
  - 1237.20.49202 Boehringer Ingelheim Investigational Site, Wiesbaden
- Hungary (5):
  - 1237.20.36202 Boehringer Ingelheim Investigational Site, Gödöllö
  - 1237.20.36204 Boehringer Ingelheim Investigational Site, Komárom
  - 1237.20.36203 Boehringer Ingelheim Investigational Site, Pécs
  - 1237.20.36201 Boehringer Ingelheim Investigational Site, Szarvas
  - 1237.20.36205 Boehringer Ingelheim Investigational Site, Százhalombatta
- Netherlands (5):
  - 1237.20.31205 Boehringer Ingelheim Investigational Site, Almelo
  - 1237.20.31202 Boehringer Ingelheim Investigational Site, Breda
  - 1237.20.31201 Boehringer Ingelheim Investigational Site, Heerlen
  - 1237.20.31204 Boehringer Ingelheim Investigational Site, Hengelo
  - 1237.20.31203 Boehringer Ingelheim Investigational Site, Zutphen

REFERENCES:
- [Derived] Beeh KM, Westerman J, Kirsten AM, Hebert J, Gronke L, Hamilton A, Tetzlaff K, Derom E. The 24-h lung-function profile of once-daily tiotropium and olodaterol fixed-dose combination in chronic obstructive pulmonary disease. Pulm Pharmacol Ther. 2015 Jun;32:53-9. doi: 10.1016/j.pupt.2015.04.002. Epub 2015 May 6. PMID 25956072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomised, double-blind, placebo-controlled, 6 treatment, 4 period, incomplete cross-over design. Each patient was randomised to one of 30 treatment sequences. Each sequence consisted of four 6-week treatment periods separated by 3-week washout periods.
Groups:
- All Subjects: Randomised, double-blind, placebo-controlled, 6 treatment, 4 period, incomplete cross-over trial to characterise the 24-hour lung function profiles of tiotropium + olodaterol fixed dose combination (2.5/5 μg, 5/5 μg), tiotropium (2.5 μg, 5 μg) and olodaterol (5 μg) (oral inhalation, delivered by the Respimat® Inhaler) after 6 weeks once daily treatment in patients with Chronic Obstructive Pulmonary Disease (COPD) [VIVACITOTM].
Period: Overall Study
Arm/Group | All Subjects
Started | 219 (Randomised)
Completed | 193 (Completed all 4 treatment periods)
Not Completed | 26
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — other than stated above | 9

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | All Subjects
Number analyzed (Participants) | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 129

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) AUC0-24h Response [L] After 6 Weeks Treatment.
Description: Area under the Forced Expiratory Volume in 1 second (FEV1) after 6 weeks treatement-time curve from 0 to 24 h post-dose, using the trapezoidal rule, divided by the duration (24 h) to report in litres.
  Mean is actually the Adjusted mean.
  The adjusted mean and standard error (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS): This patient set included patients in the Treated Set (TS) who had any period baseline and any evaluable post-dose data for the primary efficacy endpoint at any Week 6 visits.
Measure: Mean (Standard Error); unit: Litres (L)
Groups:
- Placebo: Placebo matching Tiotropium+Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT:2 Oral inhalations once daily in the morning for 6 weeks.
- Olodaterol (5 µg): Olodaterol solution for inhalation - RESPIMAT
  2 oral inhalations once daily in the morning for 6 weeks.
- Tiotropium (2.5 µg); Tiotropium (5 µg): Tiotropium solution for inhalation - RESPIMAT : 2 oral inhalations once daily in the morning for 6 weeks.
- Tiotropium+Olodaterol FDC (2.5/5 µg); Tiotropium+Olodaterol FDC (5/5 µg): Tiotropium + Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT: 2 oral inhalations once daily in the morning for 6 weeks.
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres (L) | -0.037 (0.014) | 0.129 (0.013) | 0.117 (0.013) | 0.133 (0.014) | 0.241 (0.014) | 0.244 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.280, 95% CI 2-sided [0.252 to 0.309], Standard Error of Mean 0.014 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.115, 95% CI 2-sided [0.087 to 0.143], Standard Error of Mean 0.014 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.110, 95% CI 2-sided [0.082 to 0.139], Standard Error of Mean 0.014 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.277, 95% CI 2-sided [0.249 to 0.306], Standard Error of Mean 0.015 — Adjusted mean difference to placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Median Difference (Final Values) = 0.111, 95% CI 2-sided [0.083 to 0.140], Standard Error of Mean 0.014 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.096 to 0.152], Standard Error of Mean 0.014 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Median Difference (Final Values) = 0.107, 95% CI 2-sided [0.079 to 0.136], Standard Error of Mean 0.014 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

2. Secondary Outcome: FEV1 AUC0-12h Response [L] After 6 Weeks Treatment.
Description: Area under the Forced Expiratory Volume in 1 second (FEV1) after 6 weeks treatement-time curve from 0 to 12 h post-dose, using the trapezoidal rule, divided by the duration (12h) to report in litres.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: Litres (L)
Groups:
- Placebo: Placebo matching Tiotropium+Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT: 2 Oral inhalations once daily in the morning for 6 weeks.
- Olodaterol (5 µg): Olodaterol solution for inhalation - RESPIMAT: 2 oral inhalations once daily in the morning for 6 weeks.
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres (L) | -0.013 (0.015) | 0.179 (0.015) | 0.171 (0.015) | 0.186 (0.015) | 0.310 (0.015) | 0.305 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.319, 95% CI [0.289 to 0.349], Standard Error of Mean 0.015 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.126, 95% CI 2-sided [0.096 to 0.156], Standard Error of Mean 0.015 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.119, 95% CI 2-sided [0.089 to 0.149], Standard Error of Mean 0.015 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.323, 95% CI 2-sided [0.293 to 0.354], Standard Error of Mean 0.015 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.101 to 0.161], Standard Error of Mean 0.015 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.139, 95% CI 2-sided [0.109 to 0.169], Standard Error of Mean 0.015 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.093 to 0.154], Standard Error of Mean 0.015 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

3. Secondary Outcome: FEV1 AUC12-24h Response [L] After 6 Weeks Treatment.
Description: Area under the Forced Expiratory Volume in 1 second (FEV1) after 6 weeks treatement-time curve from 12 to 24 h post-dose using the trapezoidal rule, divided by the duration (12 h) to report in litres.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres (L) | -0.060 (0.014) | 0.079 (0.013) | 0.062 (0.013) | 0.081 (0.014) | 0.172 (0.014) | 0.182 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.243, 95% CI 2-sided [0.212 to 0.273], Standard Error of Mean 0.015 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Median Difference (Final Values) = 0.103, 95% CI 2-sided [0.074 to 0.133], Standard Error of Mean 0.015 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Median Difference (Final Values) = 0.102, 95% CI 2-sided [0.072 to 0.132], Standard Error of Mean 0.015 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.232, 95% CI 2-sided [0.201 to 0.262], Standard Error of Mean 0.015 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [0.063 to 0.123], Standard Error of Mean 0.015 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.110, 95% CI 2-sided [0.080 to 0.140], Standard Error of Mean 0.015 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [0.061 to 0.121], Standard Error of Mean 0.015 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

4. Secondary Outcome: Trough FEV1 Response [L] After 6 Weeks Treatment.
Description: Trough Forced Expiratory Volume in 1 second (FEV1) response after 6 weeks treatment period.
  The trough was defined as the mean of the 23 h and 23 h50 min measurements and Response was defined as the change from patient baseline.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Litres
Groups:
- Placebo: Placebo matching Tiotropium+Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT: 2 Oral inhalations once daily in the morning for 6 weeks.)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres | -0.006 (0.015) | 0.109 (0.015) | 0.095 (0.015) | 0.122 (0.015) | 0.196 (0.015) | 0.201 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.207, 95% CI 2-sided [0.173 to 0.241], Standard Error of Mean 0.017 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.092, 95% CI 2-sided [0.059 to 0.126], Standard Error of Mean 0.017 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [0.045 to 0.113], Standard Error of Mean 0.017 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.201, 95% CI 2-sided [0.167 to 0.235], Standard Error of Mean 0.017 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.086, 95% CI 2-sided [0.052 to 0.120], Standard Error of Mean 0.017 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.067 to 0.135], Standard Error of Mean 0.017 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.073, 95% CI 2-sided [0.039 to 0.107], Standard Error of Mean 0.017 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

5. Secondary Outcome: Peak(0-3h) FEV1 Response [L] After 6 Weeks Treatment.
Description: Peak (0-3h) Forced Expiratory Volume in 1 second (FEV1) response.
  The peak was defined as the maximum value measured within the first 3 h post dosing and response was defined as the change from patient baseline.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 135 | 138 | 136 | 137 | 135 | 138
Litres (L) | 0.072 (0.017) | 0.291 (0.016) | 0.290 (0.016) | 0.300 (0.016) | 0.422 (0.016) | 0.411 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.338, 95% CI 2-sided [0.305 to 0.371], Standard Error of Mean 0.017 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.120, 95% CI 2-sided [0.087 to 0.153], Standard Error of Mean 0.017 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [0.078 to 0.143], Standard Error of Mean 0.017 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.350, 95% CI 2-sided [0.317 to 0.383], Standard Error of Mean 0.017 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.098 to 0.164], Standard Error of Mean 0.017 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.132, 95% CI 2-sided [0.099 to 0.165], Standard Error of Mean 0.017 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.122, 95% CI 2-sided [0.089 to 0.155], Standard Error of Mean 0.017 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

6. Secondary Outcome: FVC AUC0-24h Response [L] After 6 Weeks Treatment.
Description: Area under the Forced Vital Capacity (FVC) after 6 weeks treatment period-time curve from 0 to 24 h post-dose using the trapezoidal rule, divided by the duration (24 h) to report in litres.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: Litres(L)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres(L) | -0.065 (0.023) | 0.158 (0.022) | 0.172 (0.022) | 0.191 (0.022) | 0.331 (0.022) | 0.368 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.433, 95% CI 2-sided [0.389 to 0.477], Standard Error of Mean 0.022 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.210, 95% CI 2-sided [0.166 to 0.253], Standard Error of Mean 0.022 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.177, 95% CI 2-sided [0.133 to 0.221], Standard Error of Mean 0.022 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.396, 95% CI 2-sided [0.352 to 0.441], Standard Error of Mean 0.023 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.173, 95% CI 2-sided [0.129 to 0.217], Standard Error of Mean 0.022 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.159, 95% CI 2-sided [0.115 to 0.203], Standard Error of Mean 0.022 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated. is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [0.096 to 0.184], Standard Error of Mean 0.022 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

7. Secondary Outcome: FVC AUC0-12h Response [L] After 6 Weeks Treatment.
Description: Area under the Forced Vital Capacity (FVC) after 6 weeks treatment period-time curve from 0 to 12 h post-dose using the trapezoidal rule, divided by the duration (12 h) to report in litres.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres (L) | -0.023 (0.024) | 0.240 (0.024) | 0.249 (0.024) | 0.261 (0.024) | 0.420 (0.024) | 0.440 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.463, 95% CI 2-sided [0.417 to 0.509], Standard Error of Mean 0.024 — Adjusted mean difference to placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.200, 95% CI 2-sided [0.154 to 0.246], Standard Error of Mean 0.023 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.179, 95% CI 2-sided [0.133 to 0.225], Standard Error of Mean 0.023 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.443, 95% CI 2-sided [0.396 to 0.490], Standard Error of Mean 0.024 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.181, 95% CI 2-sided [0.134 to 0.227], Standard Error of Mean 0.024 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.171, 95% CI 2-sided [0.125 to 0.218], Standard Error of Mean 0.024 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.159, 95% CI 2-sided [0.113 to 0.206], Standard Error of Mean 0.024 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

8. Secondary Outcome: FVC AUC12-24h Response [L] After 6 Weeks Treatment.
Description: Area under the Forced Vital Capacity (FVC) after 6 weeks treatment period-time curve from 12 to 24 h post-dose using the trapezoidal rule, divided by the duration (12 h) to report in litres.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres (L) | -0.108 (0.023) | 0.077 (0.023) | 0.095 (0.023) | 0.122 (0.023) | 0.243 (0.023) | 0.296 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.404, 95% CI 2-sided [0.355 to 0.453], Standard Error of Mean 0.025 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.219, 95% CI 2-sided [0.170 to 0.267], Standard Error of Mean 0.025 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [0.126 to 0.223], Standard Error of Mean 0.025 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.351, 95% CI 2-sided [0.301 to 0.400], Standard Error of Mean 0.025 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.166, 95% CI 2-sided [0.117 to 0.214], Standard Error of Mean 0.025 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.148, 95% CI 2-sided [0.099 to 0.197], Standard Error of Mean 0.025 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [0.072 to 0.170], Standard Error of Mean 0.025 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

9. Secondary Outcome: Trough FVC Response [L] After 6 Weeks Treatment.
Description: Trough Forced Vital Capacity (FVC) response after 6 weeks treatment period.
  The trough was defined as the mean of the 23 h and 23 h50 min measurements and response was defined as the change from patient baseline.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day1 and week 6
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres (L) | -0.025 (0.026) | 0.134 (0.026) | 0.115 (0.026) | 0.183 (0.026) | 0.282 (0.026) | 0.304 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.329, 95% CI 2-sided [0.274 to 0.385], Standard Error of Mean 0.028 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.170, 95% CI 2-sided [0.115 to 0.225], Standard Error of Mean 0.028 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [0.066 to 0.176], Standard Error of Mean 0.028 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Median Difference (Final Values) = 0.307, 95% CI 2-sided [0.251 to 0.363], Standard Error of Mean 0.029 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.147, 95% CI 2-sided [0.092 to 0.203], Standard Error of Mean 0.028 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.166, 95% CI 2-sided [0.111 to 0.222], Standard Error of Mean 0.028 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.099, 95% CI 2-sided [0.043 to 0.154], Standard Error of Mean 0.028 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

10. Secondary Outcome: Peak (0-3h) FVC Response [L] After 6 Weeks Treatment.
Description: Peak (0-3h) Forced Vital Capacity (FVC) responses after 6 weeks treatment.
  Peak was defined as the maximum value measured within the first 3 h post dosing and response was defined as the change from patient baseline.
  Mean is actually the Adjusted mean.
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: day 1 and week 6
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Number analyzed (Participants) | 132 | 136 | 136 | 135 | 135 | 138
Litres (L) | 0.159 (0.029) | 0.463 (0.029) | 0.450 (0.029) | 0.470 (0.029) | 0.612 (0.029) | 0.621 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.462, 95% CI 2-sided [0.408 to 0.516], Standard Error of Mean 0.028 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 2: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.159, 95% CI 2-sided [0.105 to 0.212], Standard Error of Mean 0.027 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 3: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.151, 95% CI 2-sided [0.098 to 0.205], Standard Error of Mean 0.027 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated
Statistical Analysis 4: Comparison: Placebo vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.452, 95% CI 2-sided [0.398 to 0.507], Standard Error of Mean 0.028 — Adjusted mean difference to Placebo is calculated
Statistical Analysis 5: Comparison: Olodaterol (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.149, 95% CI 2-sided [0.095 to 0.203], Standard Error of Mean 0.028 — Adjusted mean difference to Olodaterol (5 µg) is calculated
Statistical Analysis 6: Comparison: Tiotropium (2.5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.161, 95% CI 2-sided [0.107 to 0.216], Standard Error of Mean 0.028 — Adjusted mean difference to Tiotropium low dose (2.5 µg) is calculated
Statistical Analysis 7: Comparison: Tiotropium (5 µg) vs Tiotropium+Olodaterol FDC (2.5/5 µg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model repeated measures (MMRM) with fixed effects for treatment,period and random effect for patient; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [0.087 to 0.196], Standard Error of Mean 0.028 — Adjusted mean difference to Tiotropium high dose (5 µg) is calculated

ADVERSE EVENTS:
Time Frame: From drug administration until 21 days after the last administration, upto 92 days.
Arm/Group | Placebo | Olodaterol (5 µg) | Tiotropium (2.5 µg) | Tiotropium (5 µg) | Tiotropium+Olodaterol FDC (2.5/5 µg) | Tiotropium+Olodaterol FDC (5/5 µg)
Serious Adverse Events (participants affected / at risk) | 4/138 | 8/138 | 5/137 | 3/138 | 4/136 | 1/139
Other Adverse Events (participants affected / at risk) | 40/138 | 21/138 | 30/137 | 29/138 | 23/136 | 25/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=138) | Olodaterol (5 µg) (N=138) | Tiotropium (2.5 µg) (N=137) | Tiotropium (5 µg) (N=138) | Tiotropium+Olodaterol FDC (2.5/5 µg) (N=136) | Tiotropium+Olodaterol FDC (5/5 µg) (N=139)
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arterial disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=138) | Olodaterol (5 µg) (N=138) | Tiotropium (2.5 µg) (N=137) | Tiotropium (5 µg) (N=138) | Tiotropium+Olodaterol FDC (2.5/5 µg) (N=136) | Tiotropium+Olodaterol FDC (5/5 µg) (N=139)
Nasopharyngitis (Infections and infestations) | 14 | 12 | 12 | 12 | 12 | 9
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 5 | 13 | 12 | 8 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 3 | 6 | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 4 | 3 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.